CLINICAL TRIAL: NCT00794820
Title: Fludarabine, Cyclophosphamide, and Multiple Dose Rituximab as Frontline Therapy in Chronic Lymphocytic Leukemia (CLL)
Brief Title: Fludarabine, Cyclophosphamide, and Rituximab - High Dose Frontline
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0591; NCI-2010-01220 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-11-18; First posted 2008-11-20 (Estimated); Results first posted 2016-08-23 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Leukemia; Fludarabine phosphate; Cyclophosphamide; Rituximab; FCR; Cytoxan®; Neosar®; Rituxan®
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — fludarabine phosphate; fludarabine; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FCR-Multiple Dose Rituximab (Experimental): Fludarabine phosphate + Cyclophosphamide + Rituximab
  Interventions: Drug: Fludarabine Phosphate; Drug: Cyclophosphamide; Drug: Rituximab

INTERVENTIONS:
Drug: Fludarabine Phosphate — 25 mg/m^2 by vein over 5-30 minutes daily for 3 days (days 2-4)
  Other Names: Fludara®; Fludarabine
Drug: Cyclophosphamide — 250 mg/m^2 by vein over 60 minutes daily for 3 days (days 2-4)
  Other Names: Cytoxan®; Neosar®
Drug: Rituximab — 375 mg/m^2 by vein for dose 1 (given 1 day prior to chemotherapy) and then 500 mg/m^2 on days 2-3
  Other Names: Rituxan®

SUMMARY:
Primary Objective:

* To evaluate the efficacy (combined morphologic and flow remissions) of a combination of fludarabine, cyclophosphamide and multiple dose rituximab as frontline therapy for CLL.

Secondary Objective:

* To evaluate remission duration and survival.

DETAILED DESCRIPTION:
DESCRIPTION OF RESEARCH

Fludarabine and cyclophosphamide are chemotherapy drugs that are used in the treatment of CLL. Rituximab is a monoclonal antibody that binds to lymphoma cells and causes cell death.

Before treatment starts, you will have a complete physical exam and routine blood tests (about 2 teaspoons). A bone marrow sample will be collected. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Women who are able to have children must have a negative blood or urine pregnancy test.

Rituximab will be given through a needle (IV) in a vein on Days 1, 2, and 3. One day after the first dose of rituximab (Day 2), fludarabine and cyclophosphamide will be given through a needle (IV) in a vein daily for 3 days (Days 2, 3, 4). After the first month, all the drugs will be given on Days 1, 2, 3. Other IV fluids such as saline will be given on all of the treatment days for hydration, which means that the daily visit will take about six hours. The combination will be repeated once every 4 to 6 weeks for a total of 6 courses.

The drugs acetaminophen (Tylenol) and diphenhydramine hydrochloride (Benadryl) will be given before the dose of rituximab. This will be done to decrease the risk of side effects. If side effects do occur during rituximab treatment, the drug may have to be stopped until the side effects go away and then restarted so the time in the outpatient area may be longer.

The first treatment will be given at M. D. Anderson. The other 5 courses can be performed ether at M. D. Anderson or at home with your regular physician.

The same doses of all three drugs will be used throughout the study unless side effects become severe. In that case, the dose may be lowered or the treatment may be stopped. You will be taken off study if the disease gets worse.

During treatments, patients will have blood samples (about 1 teaspoon each) taken once every 1-2 weeks. Bone marrow studies will be done at the end of the 3rd and 6th chemotherapy courses.

After treatment is completed, you will have blood tests (about 2 teaspoons each) done every 3 months for as long as you are in remission.

This is an investigational study. The FDA has approved all of the drugs used in this study and they are commercially available. However, their use in this study is investigational. As many as 64 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 16 years or older
2. Untreated CLL with indication for therapy or minimally treated (e.g. less than 1 month of steroids or chemotherapy) are eligible
3. Performance status of 3 or better (Appendix A)
4. Adequate renal and hepatic function (creatinine <2 mg%, bilirubin <2mg%). Patient with renal or liver dysfunction due to organ infiltration by lymphocytes may be eligible after discussion with the study chairman but upper limits for creatinine even under these circumstances would be creatinine < 3 mg% and bilirubin < 6 mg%. Patients with Gilbert's Syndrome may be entered on study with bilirubin 2-7 mg%..
5. A signed informed consent in keeping with policies of the hospital

Exclusion Criteria:

1) None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2003-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan O'Brien, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- FCR-Multiple Dose Rituximab: Fludarabine phosphate 25 mg/m^2 intravenous (IV) daily for 3 days (days 2-4) + Cyclophosphamide 250 mg/m^2 IV daily for 3 days (days 2-4)+ Rituximab 375 mg/m^2 IV for dose 1 (given 1 day prior to chemotherapy) then 500 mg/m^2 on days 2-3
Period: Overall Study
Arm/Group | FCR-Multiple Dose Rituximab
Started | 66
Completed | 50
Not Completed | 16
Not completed — Adverse Event | 11
Not completed — Secondary Malignancies | 2
Not completed — Resistant Disease | 2
Not completed — Ineligible/Screen Failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | FCR-Multiple Dose Rituximab
Number analyzed (Participants) | 66
Age, Continuous [Median (Full Range); unit: years] | 58 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 53
Region of Enrollment [Number; unit: participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate of FCR3 in Treatment-naïve Participants With Chronic Lymphocytic Leukemia (CLL) at 6 Months
Description: CR Rate is defined as number of all treated participants with CR as defined by 2008 IWCLL update of NCI-WG response criteria: Complete remission (CR), requiring absence of peripheral blood clonal lymphocytes by immunophenotyping, absence of lymphadenopathy, absence of hepatomegaly or splenomegaly, absence of constitutional symptoms and satisfactory blood counts; Complete remission with incomplete marrow recovery (CRi), defined as CR above, but without normal blood counts; Partial remission (PR), defined as ≥ 50% fall in lymphocyte count, ≥ 50% reduction in lymphadenopathy or ≥ 50% reduction in liver or spleen, together with improvement in peripheral blood counts; Progressive disease (PD): ≥ 50% rise in lymphocyte count to > 5 x109/L, ≥ 50% increase in lymphadenopathy, ≥ 50% increase in liver or spleen size, Richter's transformation, or new cytopenias due to CLL; Stable disease, defined as not meeting criteria for CR, CRi, PR or PD.
Time Frame: 6 months
Population: Of the 66 participants registered, one participant failed screening and therefore was not evaluable for toxicity or response. One of the 65 participants was not assessed for response to therapy therefore is not included in analysis. The participant went off study after two months of treatment and was not evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | FCR-Multiple Dose Rituximab
Number analyzed (Participants) | 64
Percentage of Participants | 75

2. Secondary Outcome: Remission Duration/Time to Progression (TTP)
Description: TTP was defined as time from initiation of treatment to primary refractory disease or CLL progression. TTP was censored for therapy-related myelodysplastic syndrome (t-MDS) or acute myelogenous leukemia (t-AML) and death in remission. TTP calculated using Kaplan-Meier estimates.
Time Frame: 6 months to disease progression, period covered up to 12 years following treatment; Data cutoff for analysis was October 2014.
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | FCR-Multiple Dose Rituximab
Number analyzed (Participants) | 64
Months | 81 [1 to 130]

3. Secondary Outcome: Overall Survival (OS) Rate
Description: OS was defined as the time from the initiation of treatment to last follow-up date or death. OS were calculated using Kaplan-Meier estimates.
Time Frame: as for outcome 2
Population: Of the 66 participants registered, one participant failed screening and therefore was not evaluable for toxicity or response. One of the 65 participants is not included in analysis, the participant went off study after two months of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | FCR-Multiple Dose Rituximab
Number analyzed (Participants) | 64
Percentage of Participants | 58

ADVERSE EVENTS:
Time Frame: Adverse events collected through 6 courses; courses repeated every 4-6 weeks, up to 36 weeks.
Description: Of the 66 participants registered, one participant failed screening and therefore was not evaluable for toxicity or response.
Arm/Group | FCR-Multiple Dose Rituximab
Serious Adverse Events (participants affected / at risk) | 30/65
Other Adverse Events (participants affected / at risk) | 63/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCR-Multiple Dose Rituximab (N=65)
Infection (Infections and infestations) | 24 (31)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Pain (General disorders) | 2 (2)
Bacteria Infection (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCR-Multiple Dose Rituximab (N=65)
Nausea (Gastrointestinal disorders) | 46 (97)
Vomiting (Gastrointestinal disorders) | 6 (7)
Fatigue (General disorders) | 42 (68)
Diarrhea (Gastrointestinal disorders) | 8 (11)
Rash (Skin and subcutaneous tissue disorders) | 7 (8)
Edema (General disorders) | 7 (9)
Fever (General disorders) | 41 (66)
Chills (General disorders) | 21 (25)
Pain (General disorders) | 18 (25)
Other Infection (Infections and infestations) | 4 (4)
Thromboembolic event (Vascular disorders) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 7 (8)
Neutropenia (Blood and lymphatic system disorders) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes